CLINICAL TRIAL: NCT05135663
Title: A Phase II, Open-Label, Extension Study of NS-089/NCNP-02 in Patients With Duchenne Muscular Dystrophy
Brief Title: Extension Study of NS-089/NCNP-02 in DMD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS089/NCNP02-P2OE; jRCT2031210162 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-10-05; First posted 2021-11-26 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NS-089/NCNP-02 40 mg/kg (Experimental)
  Interventions: Drug: NS-089/NCNP-02
- NS-089/NCNP-02 80 mg/kg (Experimental)
  Interventions: Drug: NS-089/NCNP-02

INTERVENTIONS:
Drug: NS-089/NCNP-02 — The same dose administered in as Part 2 of Study NCNP/DMT02 (40 mg/kg) will be administered once weekly for 288 weeks (The total treatment period is 312 weeks including Part2 of Study NCNP/DMT02).
  Other Names: Brogidirsen
  Arms: NS-089/NCNP-02 40 mg/kg
Drug: NS-089/NCNP-02 — The same dose administered in as Part 2 of Study NCNP/DMT02 (80 mg/kg) will be administered once weekly for 288 weeks (The total treatment period is 312 weeks including Part2 of Study NCNP/DMT02).
  Other Names: Brogidirsen
  Arms: NS-089/NCNP-02 80 mg/kg

SUMMARY:
This is the extension study of NS-089/NCNP-02 (Study NCNP/DMT02), which is designed to assess the safety, tolerability and efficacy of NS-089/NCNP-02 in patients with Duchenne muscular dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

1. Patient completed Study NCNP/DMT02

Exclusion Criteria:

1. Patient had any serious adverse events in Study NCNP/DMT02 that, in the opinion of the Investigator and/or Sponsor, was probably or definitely related to NS-089/NCNP-02 use and precludes safe use of NS-089/NCNP-02 for the patient in this study.
2. Patient had a treatment which was made for the purpose of dystrophin or dystrophin-related protein induction after completion of Study NCNP/DMT02.
3. Patient took any other investigational drugs after completion of Study NCNP/DMT02.
4. Patient was judged by the investigator and/or the Sponsor that it was not appropriate to participate in the extension study for other reasons.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to Week 319

SECONDARY OUTCOMES:
Expression of dystrophin protein (Western blot) | Week 99
Percentage of exon 44-skipped mRNA of dystrophin | Week 99
North Star Ambulatory Assessment (NSAA) | Up to Week 315
Time to stand test | Up to Week 315
Time to run/walk 10 meters test | Up to Week 315
Six-minute walk test/Two-minute walk test | Up to Week 315
Timed Up & Go test | Up to Week 315
Quantitative muscle strength assessment | Up to Week 315
Performance of Upper Limb test | Up to Week 315
Change in serum creatine kinase concentration from baseline | Up to Week 315

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Kagoshima University Hospital, Kagoshima
  - National Center of Neurology and Psychiatry, Tokyo